CLINICAL TRIAL: NCT05142436
Title: BAT3221032: A Randomized, Controlled Study to Evaluate the Effects of Switching From Cigarette Smoking to Using One of Five Variants of a Heated Tobacco Product on Biomarkers of Exposure and Biomarkers of Potential Harm in Healthy Subjects
Brief Title: BAT3221032: A Study to Evaluate the Effects of Switching From Cigarette Smoking to Using One of Five Variants of a Heated Tobacco Product on Biomarkers of Exposure and Biomarkers of Potential Harm in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British American Tobacco (Investments) Limited (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BAT3221032
Record Dates: First submitted 2021-11-16; First posted 2021-12-02 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Smoking; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort 1: Non-combusted cigarette variant 42001402 and product use mode B (Experimental): Subjects randomized to use of a non-combusted cigarette variant and product use mode B
  Interventions: Other: Product A: Non-Combusted Cigarette Variant 42001402 and product use Mode B
- Cohort 2: Non-combusted cigarette variant 42001399 and product use mode B (Experimental): Subjects randomized to use of a non-combusted cigarette variant and product use mode B
  Interventions: Other: Product B: Non-Combusted Cigarette Variant 42001399 and product use Mode B
- Cohort 3: Non-combusted cigarette variant 42001401 and product use mode B (Experimental): Subjects randomized to use of a non-combusted cigarette variant and product use mode B
  Interventions: Other: Product C: Non-Combusted Cigarette Variant 42001401 and product use Mode B
- Cohort 4: Non-combusted cigarette variant 40007386 and product use mode B (Experimental): Subjects randomized to use of a non-combusted cigarette variant and product use mode B
  Interventions: Other: Product D: Non-Combusted Cigarette Variant 40007386 and product use Mode B
- Cohort 5: Non-combusted cigarette variant 42001402 and product use mode A (Experimental): Subjects randomized to use of a non-combusted cigarette variant and product use mode A
  Interventions: Other: Product E: Non-Combusted Cigarette Variant 42001402 and product use Mode A
- Cohort 6: Usual Brand Cigarettes (No Intervention): Subjects randomized to continue to smoke usual brand cigarettes
- Cohort 7: Assisted Smoking Cessation (No Intervention): Subjects assigned to assisted smoking cessation
- Cohort 8: Never-Smokers (No Intervention): Never-smokers

INTERVENTIONS:
Other: Product A: Non-Combusted Cigarette Variant 42001402 and product use Mode B — 42001402, A Heated Tobacco Product using a Non-Combusted Cigarette Variant and product use Mode B
  Arms: Cohort 1: Non-combusted cigarette variant 42001402 and product use mode B
Other: Product B: Non-Combusted Cigarette Variant 42001399 and product use Mode B — 42001399, A Heated Tobacco Product using a Non-Combusted Cigarette Variant and product use Mode B
  Arms: Cohort 2: Non-combusted cigarette variant 42001399 and product use mode B
Other: Product C: Non-Combusted Cigarette Variant 42001401 and product use Mode B — 42001401, A Heated Tobacco Product using a Non-Combusted Cigarette Variant and product use Mode B
  Arms: Cohort 3: Non-combusted cigarette variant 42001401 and product use mode B
Other: Product D: Non-Combusted Cigarette Variant 40007386 and product use Mode B — 40007386, A Heated Tobacco Product using a Non-Combusted Cigarette Variant and product use Mode B
  Arms: Cohort 4: Non-combusted cigarette variant 40007386 and product use mode B
Other: Product E: Non-Combusted Cigarette Variant 42001402 and product use Mode A — 42001402, A Heated Tobacco Product using a Non-Combusted Cigarette Variant and product use Mode A
  Arms: Cohort 5: Non-combusted cigarette variant 42001402 and product use mode A

SUMMARY:
This is a randomized, controlled, multi-center, open-label, 8-cohort parallel group study to assess changes in select biomarkers of exposure (BoE) and biomarkers of potential harm (BoPH) in generally healthy smokers switching to the study investigational products (IPs), compared to subjects who continue to smoke, undergo smoking abstinence, or have never smoked.

DETAILED DESCRIPTION:
All subjects will participate in a baseline biomarker assessment and smokers will then be switched to exclusive use of their assigned product (cohorts 1-5), continue to smoke (cohort 6), or smoking cessation (cohort 7), and never-smokers will continue to not smoke (cohort 8). Subjects will be directed to use their assigned product exclusively for 3 months and will participate in study visits throughout the study for safety, product re-supply and collection of samples for biomarker assessments. Throughout the study, subjects will report their daily use of the study IP and/or cigarette smoking.

This study will be ambulatory, with subjects in cohorts 1-7 attending a total of 4 clinic visits (one every approximately 30 days) over a period of 3 months. Subjects in cohorts 1-7 will be confined in the study site overnight the night before their Day 1 (Visit 1, baseline) and Day 90 (Visit 4) visits. The Day 30 (Visit 2) and Day 60 (Visit 3) visits will be non-residential visits for pregnancy testing (female subjects) and product usage assessments and resupply only. Subjects in cohort 8 will attend the clinic for Visit 1 and Visit 4 only, and will be confined in the clinic overnight the night before each of these visits. In addition, all subjects will attend a Screening Visit.

Smokers will be asked to continue smoking their usual brand (UB) cigarettes until randomization (cohorts 1-6) or enrollment (cohort 7) at Visit 1. Never-smokers will be asked to continue not to use any tobacco or nicotine products for the entire study duration.

All subjects will be confined on Visit 1 and will use their UB cigarettes ad libitum during this period (unless required to abstain for specific tests and excluding cohort 8, who will not use any nicotine or tobacco products). Exhaled breath, 24-hour urine and blood samples will be collected and evaluated for baseline BoE and BoPH. Smokers of non-menthol UB cigarettes will then be randomized to cohort 1, 5 or 6; smokers of mentholated UB cigarettes will be randomized to cohort 2, 3, 4 or 6; smokers who intend to quit smoking will be enrolled to cohort 7; and never-smokers will be enrolled to cohort 8.

All subjects will be confined on Visit 4. Subjects in cohorts 1-6 will use their assigned product exclusively, ad libitum during this period (unless required to abstain for specific tests). Other than subjects in cohort 7 who are using nicotine replacement therapy as part of their smoking cessation strategy, subjects in cohorts 7 and 8 will not use any tobacco or nicotine products. Exhaled breath, 24-hour urine and blood samples will be collected and evaluated for BoE and BoPH.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English or Spanish.
2. Generally healthy male or female, 26 to 55 years of age, inclusive, at the time of consent.
3. Body mass index (BMI) within 18.0 to 40.0 kg/m2, inclusive (minimum weight of at least 110 lbs. [50 kg]) at Screening.
4. Agree to abide by the study restrictions and requirements, including use of the assigned product or to undergo smoking cessation, and agree to in-clinic, overnight confinement at Visits 1 and 4.
5. Willing to refrain from consuming alcohol within 24 hours prior to Screening and check-in at Visits 1 and 4.
6. Willing to refrain from consuming cruciferous vegetables and grilled, smoked, fried or barbequed food, and to avoid being in the presence of the cooking of these foods, and to refrain from consuming cured sandwich meats, bacon, salami, and sausages, for 48 hours prior to check-in at Visits 1 and 4.
7. Males must be vasectomized, abstinent from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation), or they (or their female partner of childbearing potential) must use acceptable methods of birth control from Visit 1 until the end of the study.
8. Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until the end of the study.

   Examples of acceptable means of birth control are, but not limited to:
   1. Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy);
   2. Established use of oral, implantable, injectable or transdermal methods of contraception associated with inhibition of ovulation;
   3. Physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide;
   4. Non-hormone releasing intrauterine devices (IUD) or hormone-releasing IUDs (e.g., Mirena or Kyleena);
   5. Vasectomized partner;
   6. Abstinence from heterosexual intercourse (as a lifestyle choice, not just for the purpose of study participation); and
   7. Post-menopausal and not on hormone replacement therapy.

   Cohorts 1 to 7
9. Smokes manufactured combustible, filtered, non-menthol (cohorts 1 and 5) or menthol (cohorts 2, 3 and 4) cigarettes (either is acceptable for cohorts 6 and 7), 83 mm to 100 mm in length as their primary source of nicotine.
10. Has smoked for at least the five consecutive years prior to Screening. Brief periods of abstinence due to illness, quit attempt (more than 30 days prior to Screening), or clinical study participation (more than 30 days prior to Screening) will be allowed at the discretion of the PI.
11. Smokes an average of at least 10 and a maximum of 30 cigarettes per day (CPD) and inhales the smoke.
12. Exhaled breath carbon monoxide (eCO) level is ≥ 7 ppm and ≤ 100 ppm at Screening.
13. Positive urine cotinine test at Screening.
14. If assigned to cohort 1, 2, 3, 4 or 5, willing to use only the study product (HTP) provided to them during the study.
15. If assigned to cohort 6, willing to continue to smoke factory-manufactured cigarettes.
16. For cohort 7 only, willing to refrain from smoking or using any form of tobacco or nicotine-containing product (other than nicotine replacement therapy (NRT) where agreed as part of their smoking cessation strategy).
17. Agree not to allow any other person to use any product provided to them for use during this study, nor to dispose of any product provided to them for use during this study with the exception of the disposal of used HTP sticks or used NRT.

    Cohort 8
18. Never have smoked (<100 cigarettes in their life), not have smoked or used any nicotine or tobacco product within 30 days prior to Screening, and will continue not to smoke or use any form of tobacco or nicotine-containing product (including HTPs) for the duration of the study.
19. Lives in a non-smoking household and is not employed in a role which regularly exposes them to tobacco smoke (e.g., bar worker).
20. Exhaled breath carbon monoxide (eCO) level is < 7 ppm at Screening.
21. Negative urine cotinine test at Screening.

Exclusion Criteria:

All Subjects

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease(s), or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes (history of gestational diabetes which is no longer present nor indicated by clinical laboratory test results is acceptable).
3. Treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
4. Subjects who have had an acute illness (e.g., upper respiratory tract infection) requiring treatment within 4 weeks prior to Visit 1 (subjects who had viral infections that resolved ≥ 2 weeks prior to Visit 1 will be admissible).
5. Subjects who have received any medications or substances (other than nicotine) which:

   1. interfere with the cyclooxygenase pathway (e.g., anti-inflammatory drugs including aspirin and ibuprofen) within 14 days prior to Visit 1
   2. are known to be strong inducers or inhibitors of cytochrome P450 (CYP) enzymes within 14 days or 5 half-lives of the drug (whichever is longer) prior to Visit 1
6. History or presence of bleeding or clotting disorders.
7. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
8. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes.
9. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
10. Positive urine/saliva drug screen without evidence of prescribed corresponding concomitant medication(s) at the Screening Visit or Visit 1, with the exception of for tetrahydrocannabinol (THC). If positive for THC, a cannabis intoxication evaluation will be performed at check-in, and inclusion will be at the discretion of the PI or appropriately qualified designee.
11. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
12. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
13. Participation in another clinical trial within (≤) 30 days prior to signing the ICF. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing informed consent in the current study.
14. Subjects who have donated:

    1. ≥400 mL of blood within 30 days prior to screening, or during the period from signing informed consent to check-in at Visit 1
    2. plasma in the 7 days prior to screening, or during the period from signing informed consent to the end of study (Visit 4)
15. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
16. Has a significant history of alcoholism or drug abuse within 24 months prior to Screening, as determined by the PI, or has a positive urine/breath alcohol test at Screening or Visit 1.
17. Determined by the PI to be inappropriate for this study.

    Cohorts 1 to 6
18. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous attempt within 30 days prior to the signing of the ICF.
19. Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to the signing the ICF.

    Cohorts 1 to 7
20. Currently uses any nicotine or tobacco product, other than CC, more than one day per week.

Ages: 26 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 806 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Total NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol [NNAL] + glucuronides) | 90 days
  To quantitively assess differences in biomarker of exposure, Total NNAL, at 90 days between subjects who continue to smoke combustible cigarettes (CC) and subjects who switch to an HTP
Monohydroxybutyl mercapturic acid (MHBMA) | 90 days
  To quantitively assess differences in biomarker of exposure, MHBMA, at 90 days between subjects who continue to smoke CC and subjects who switch to an HTP
3-hydroxypropyl mercapturic acid (3-HPMA) | 90 days
  To quantitively assess differences in biomarker of exposure, 3-HPMA, at 90 days between subjects who continue to smoke CC and subjects who switch to an HTP
S-phenyl mercapturic acid (S-PMA) | 90 days
  To quantitively assess differences in biomarker of exposure, S-PMA, at 90 days between subjects who continue to smoke CC and subjects who switch to an HTP
Carboxyhemoglobin (COHb) | 90 days
  To quantitively assess differences in biomarker of exposure, COHb, at 90 days between subjects who continue to smoke CC and subjects who switch to an HTP

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Gale, Study Director — BAT
Locations (18):
- United States (18):
  - Pillar Clinical Research, LLC, Bentonville, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, Rogers, Arkansas
  - Bright Research Center, Miami, Florida
  - Infinite Clinical Trials, Morrow, Georgia
  - AMR Lexington, Lexington, Kentucky
  - AMR Kansas City, Kansas City, Missouri
  - QPS Bio-Kinetic, Springfield, Missouri
  - High Point Clinical Trials Center, High Point, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Centricity Research, Columbus, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - AMR Knoxville, Knoxville, Tennessee
  - InSite Clinical Research, LLC., DeSoto, Texas
  - Pillar Clinical Research, Richardson, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No